CLINICAL TRIAL: NCT05475522
Title: Intraoperative Sonographically Guided Versus 5-Aminolevulinic Acid Fluorescence Guided Resection of Gliomas and Brain Metastases Enhancing Contrast Agent in Magnetic Resonance Imaging: a Randomised, Controlled, Noninferiority Trial
Brief Title: Intraoperative Sonographically Versus Fluorescence-guided Resection of Contrast-enhancing Gliomas and Brain Metastases
Acronym: SONOFLUO
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: technical issues
Sponsor: Sklifosovsky Institute of Emergency Care (Other Government)
Responsible Party: Principal Investigator, Alexander Dmitriev, Principal Investigator, Sklifosovsky Institute of Emergency Care
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 9b
Record Dates: First submitted 2022-07-22; First posted 2022-07-27 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Gliomas, Malignant; Metastases to Brain
Keywords: contrast-enhancing glioma; brain metastasis; sonography; ultrasound; fluorescence; 5-aminolevulinic acid; 5-ALA
MeSH Terms: conditions — Glioma; Brain Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Tumor extent of resection will be assessed by radiologists blinded for the treatment arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ultrasound (Experimental): Intraoperative extent of tumor resection will be assessed using sonography
  Interventions: Device: Ultrasound guided brain tumor resection
- Fluorescence (Active Comparator): Intraoperative extent of tumor resection will be assessed using fluorescence with 5-aminolevulinic acid
  Interventions: Device: 5-aminolevulinic acid fluorescence-guided brain tumor resection

INTERVENTIONS:
Device: Ultrasound guided brain tumor resection — Surgeon intraoperatively assesses extent of tumor resection using ultrasound
  Arms: Ultrasound
Device: 5-aminolevulinic acid fluorescence-guided brain tumor resection — Surgeon intraoperatively assesses extent of tumor resection observing it's fluorescence in microscope
  Arms: Fluorescence

SUMMARY:
Objective of the study is to determine whether intraoperative ultrasound guided resection of gliomas with contrast enhancement in magnetic resonance imaging and brain metastases can achieve as high rate of gross total resection as fluorescence-guided surgery with 5-aminolevulinic acid

DETAILED DESCRIPTION:
Fluorescence with 5-aminolevulinic acid, fluorescein and intraoperative magnetic resonance imaging (MRI) are the most common modalities used to intraoperatively rate extent of brain tumor resection. Intraoperative sonography is another promising method of intraoperative visualization. It's advantages include possibility of real-time estimation of tumor remnants without disturbing of surgical workflow, opportunity to discover residual tumor under normal brain tissue and chipper cost. At this time there are no published results of randomized control trials comparing ultrasound and fluorescence-guided brain tumor resection.

Objective of this study is to determine whether intraoperative ultrasound guided resection of gliomas with contrast enhancement in magnetic resonance imaging and brain metastases can achieve as high rate of gross total resection as 5-aminolevulinic acid fluorescence-guided surgery.

Participants of the study will be randomly operated using intraoperative ultrasound or fluorescence with 5-aminolevulinic acid. Extent of resection will be assessed in postoperative MRI by blinded radiologists

ELIGIBILITY:
Inclusion Criteria:

* single gliomas with contrast enhancement in preoperative magnetic resonance imaging (presumed high-grade gliomas)
* one or several brain metastases
* newly diagnosed
* Karnofsky Performance Status 60-100%
* age 18-79 years
* performed magnetic resonance imaging with contrast enhancement

Exclusion Criteria:

* tumor spreading to corpus callosum or brainstem
* previously performed brain radiotherapy
* planned supratotal tumor resection until neurophysiologically revealed eloquent areas
* known hypersensibility to 5-aminolevulinic or to porphyrin
* hepatic or renal insufficiency
* porphyria
* pregnancy
* breast feeding

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Gross total resection (Yes or No) | within 48 hours after surgery
  No residual contrast enhancement in postoperative T1-weighted magnetic resonance imaging

SECONDARY OUTCOMES:
Extent of resection (in percents) | within 48 hours after surgery
  Extent of resection = (preoperative tumor volume - postoperative tumor volume) / preoperative tumor volume x 100
Motor function (in grades) | within 10 days after surgery
  Motor function is assessed in Medical Research Council scale
Speech function (in grades) | within 10 days after surgery
  Speech function is assessed in Hendrix scale (2017)
Karnofsky performance status (in percents) | within 10 days after surgery
  Assesses patients' possibilities to self-service in Karnofsky Performance Status scale
Cerebral complications | From admission to intensive care unit after surgery till hospital discharge, up to 365 days
  Which cerebral complications arose after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Dmitriev, MD, Principal Investigator — Sklifosovsky Institute of Emergency Care
Locations (1):
- Sklifosovsky Institute of Emergency Care, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No